CLINICAL TRIAL: NCT03727373
Title: Qualitative Study for Pain Measurement Using Innovative Health Technology (QualiPain)
Brief Title: Qualitative Study for Pain Measurement Using Innovative Health Technology
Acronym: QualiPain
Status: Completed | Type: Observational
Sponsor: University Hospital Schleswig-Holstein (Other)
Collaborators: European Regional Development Fund (Other); Zealand University Hospital (Other); Design School Kolding (Other)
Responsible Party: Principal Investigator, Prof. Dirk Rades, MD, Professor Dr. med., University Hospital Schleswig-Holstein
Other Study IDs: QualiPain
Record Dates: First submitted 2018-10-30; First posted 2018-11-01 (Actual); Results first posted 2020-03-27 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Pain Measurement; Pain, Chronic; Pain, Acute; Pain, Cancer
Keywords: Pain measurement; Pain, Chronic or acute; Pain, Cancer; Health technology
MeSH Terms: conditions — Chronic Pain; Acute Pain; Cancer Pain; Pain; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The present study is a multicenter, explorative, qualitative study. The primary endpoint of this study is to evaluate to which extent the collection of data with regard to pain caused by illness or treatment can be optimized using health technology solutions. For this evaluation semi-structured qualitative interviews with 8-10 patients will be conducted.

Secondary variables are the evaluation of the patients' pain experience and the general patients' willingness to collect data with regard to pain by using technological devices themselves or with support of healthcare professionals.

DETAILED DESCRIPTION:
The present multicenter study is an explorative, qualitative study. It shall be evaluated from the patients' point of view if and how the collection of data with regard to pain, caused by illness or treatment, can be optimized using health technology solutions. A health technology solution could for example be an app for registering the intensity and localization of pain. The aim of this study is to examine, if such a solution would be accepted by patients with acute or chronic pain and how a fitting solution should be designed to meet the patients' requirements. Existing methods for pain measurement as well as possibilities for the development of new methods will be examined and evaluated during the interviews.

To arguable this issue the interviews comprise different topics like:

* the patients pain experience in everyday life, e.g. how the patients cope with pain in everyday life and how and if this is documented;
* experiences with and the thought of regular pain recording;
* an evaluation if patients tend to be willing to record their pain using technological devices by themselves or rather with support of healthcare professionals.

It is the aim to use the results of this study for the development of a new and improved version of pain registration. The results of the study will be summarized in a report and handed over to a startup company. Thereupon the startup company has the possibility to develop a technological solution that represents the patients' need at its best.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Pain intensity > 4 (numeric ranking scale 0-10)
* Legal capacity
* Written informed consent

Exclusion Criteria:

* Lack of willingness to cooperate
* Lack of consent
* Lack of ability to follow instructions
* younger than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — It is intended to have a balanced inclusion of at least 3 male and 3 female patients.
Study Population: Male and female patients with chronic or actue pain caused by illness or treatment. This pain has to be 4 or higher on a numeric ranking scale (0-10).
  The inclusion of patients is planned according to the following sample design:
  * Gender: male=3 patients; female=3 patients;
  * Age: 18-49 years = 1 patient; 50-79 years = 1 patient; >80 years = 1 patient
  * Quality of pain: acute: 2 patients; chronic: 2 patients
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2018-10-17 (Actual); Primary Completion 2018-11-23 (Actual); Study Completion 2018-11-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Rades, Prof. Dr., Principal Investigator — Dep. of Radiation Oncology, Univ. Medical Center S-H Campus Lübeck (Germany)
Locations (2):
- Germany (2):
  - Department of Neurosurgery, University Medical Center Schleswig-Holstein Campus Lübeck, Lübeck, Schleswig-Holstein
  - Department of Radiation Oncology, University of Lübeck and University Medical Center Schleswig-Holstein, Lübeck

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wilkie DJ, Judge MK, Berry DL, Dell J, Zong S, Gilespie R. Usability of a computerized PAINReportIt in the general public with pain and people with cancer pain. J Pain Symptom Manage. 2003 Mar;25(3):213-24. doi: 10.1016/s0885-3924(02)00638-3. PMID 12614956
- [Background] Tong A, Sainsbury P, Craig J. Consolidated criteria for reporting qualitative research (COREQ): a 32-item checklist for interviews and focus groups. Int J Qual Health Care. 2007 Dec;19(6):349-57. doi: 10.1093/intqhc/mzm042. Epub 2007 Sep 14. PMID 17872937
- [Background] Jaatun, A. A. E. & M. G. Jaatun. 2016. Advanced Healthcare Services Enabled by a Computerized Pain Body Map. The 6th International Conference on Current and Future Trends of Information and Communication Technologies in Healthcare (ICTH 2016).
- [Background] Kvale, S. & Brinkmann, S. 2009. Interview: Introduktion til et håndværk. Hans Reitzel Kbh.
- [Background] Rubow, Cecilie. 2003. Samtalen som deltagerobservation. In: Ind i Verden. En Grundbog i Antropologisk Metode.

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients With Acute or Chronic Pain: Patients included in this study must have had acute or chronic pain with an intensity of >4 on a numeric self-rating scale ranging from 0 to 10 (0=no pain, 10=maximum pain).
Period: Overall Study
Arm/Group | Patients With Acute or Chronic Pain
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients With Acute or Chronic Pain
Number analyzed (Participants) | 8
Age, Customized [Median (Full Range); unit: years]
  Age | 62 [31 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 8
Region of Enrollment [Number; unit: participants]
  Germany | 8
Type of pain [Count of Participants; unit: Participants]
  Acute pain | 4
  Chronic pain | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Willing to Assess Their Pain Using Technology
Description: Patients were asked during a semi-structured qualitative interview, if they were willing to assess their pain using technology.
Time Frame: 1 day (during the interview)
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Acute or Chronic Pain
Number analyzed (Participants) | 8
Participants
  Willing to assess pain using technology | 5
  Not willing to assess pain using technology | 3

2. Secondary Outcome: Number of Participants Impaired by Pain During Daily Life
Description: Patients were asked during a semi-structured qualitative interview, if they were impaired by pain during their daily life.
Time Frame: 1 day (during the interview)
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Acute or Chronic Pain
Number analyzed (Participants) | 8
Participants
  Impaired by pain during daily life | 7
  Not impaired by pain during daily life | 1

3. Secondary Outcome: Number of Participants Satisfied With Assessment of Pain Performed by Medical Staff Members
Description: Patients were asked during a semi-structured qualitative interview, if they were satisfied with the assessment of their pain when performed by medical staff members.
Time Frame: 1 day (during the interview)
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Acute or Chronic Pain
Number analyzed (Participants) | 8
Participants
  Satisfied with pain-assessment by medical staff | 5
  Not satisfied with pain-assessment by med. staff | 3

4. Secondary Outcome: Number of Participants Considering Regular Assessment of Pain Important
Description: Patients were asked during a semi-structured qualitative interview, if they were considering regular assessment of their pain important.
Time Frame: 1 day (during the interview)
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Acute or Chronic Pain
Number analyzed (Participants) | 8
Participants
  Considering regular pain-assessment important | 4
  Not considering regular pain-assessment important | 4

5. Secondary Outcome: Number of Participants Already Using Technology for Assessment of Pain or Other Medical Symptoms/Outcomes (e.g. Blood Pressure)
Description: Patients were asked during a semi-structured qualitative interview, if they were already using technology for assessment of pain or other medical symptoms/outcomes (e.g. blood pressure).
Time Frame: 1 day (during the interview)
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Acute or Chronic Pain
Number analyzed (Participants) | 8
Participants
  Already using technology | 7
  Not already using technology | 1

6. Secondary Outcome: Number of Participants Willing to Assess Their Pain Themselves
Description: Patients were asked during a semi-structured qualitative interview, if they were willing to assess their pain themselves.
Time Frame: 1 day (during the interview)
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Acute or Chronic Pain
Number analyzed (Participants) | 8
Participants
  Willing to assess pain themselves | 4
  Not willing to assess pain themselves | 4

7. Secondary Outcome: Number of Participants Willing to Assess Their Pain Using Technology, if Required by Treating Physician
Description: Patients were asked during a semi-structured qualitative interview, if they were willing to assess their pain using technology, if required by their treating physician.
Time Frame: 1 day (during the interview)
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Acute or Chronic Pain
Number analyzed (Participants) | 8
Participants
  Willing to use technology (required by physician) | 5
  Not willing to use technology (requ. by physician) | 3

8. Secondary Outcome: Number of Participants Willing to Assess Their Pain Using Technology for Their Own Interest Only
Description: Patients were asked during a semi-structured qualitative interview, if they were willing to assess their pain using technology, if this was for their own interest only.
Time Frame: 1 day (during the interview)
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Acute or Chronic Pain
Number analyzed (Participants) | 8
Participants
  Willing to use technology (own interest only) | 2
  Not willing to use technology (own interest only) | 6

ADVERSE EVENTS:
Time Frame: 1 day (day of the interview)
Arm/Group | Patients With Acute or Chronic Pain
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-09-29): https://cdn.clinicaltrials.gov/large-docs/73/NCT03727373/Prot_SAP_000.pdf
  • Informed Consent Form (2018-07-30): https://cdn.clinicaltrials.gov/large-docs/73/NCT03727373/ICF_001.pdf